CLINICAL TRIAL: NCT03898531
Title: Mineral-Nano-Pathology : Wear of Hip Implants
Brief Title: Mineral Nano Pathology
Acronym: MINAPUIH
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: MINAPATH Développement (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0623; 2018-A03343-52 (Other: ANSM)
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Arthroplasty
Keywords: hip arthroplasty; hip prosthesis resection; first implantation; wear particles
MeSH Terms: interventions — Polyethylene; Metals; Ceramics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * The synovial fluid is removed by syringe during the surgery,
  * the resected synovial membrane is retrieved,
  * the femoral head or components removed from the prosthesis are retrieved,
  * routine biological sampling is performed during surgery to assess the patient's infectious condition
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- hip prosthesis metal/polyethylene in simple mobility
  Interventions: Procedure: hip prosthesis removed metal / polyethylene, simple mobility
- hip prosthesis metal/polyethylene in double mobility
  Interventions: Procedure: hip prosthesis removed metal / polyethylene, double mobility
- hip prosthesis ceramic/polyethylene in simple mobility
  Interventions: Procedure: hip prosthesis removed ceramic/ polyethylene, simple mobility
- hip prosthesis ceramic/polyethylene in double mobility
  Interventions: Procedure: hip prosthesis removed ceramic/ polyethylene, double mobility
- Primary implanted hip prosthesis
  Interventions: Procedure: Primary implanted hip prosthesis
- metal / metal prosthesis removed
  Interventions: Procedure: hip prosthesis removed metal/metal
- ceramic / ceramic prosthesis removed
  Interventions: Procedure: hip prosthesis removed ceramic/ceramic

INTERVENTIONS:
Procedure: hip prosthesis removed metal / polyethylene, simple mobility — Patients are hospitalized in order to change their hip prosthesis at the hospital "la Croix-Rousse" in Lyon.
  Patients have to complete before the surgery a survey on occupational and environmental exposures to mineral dust.
  The prosthesis removed is composed by metal/polyethylene. It's a simple mobility The aim is to define the types of particles that cause the most tissue inflammation
  Groups: hip prosthesis metal/polyethylene in simple mobility
Procedure: hip prosthesis removed metal / polyethylene, double mobility — Patients are hospitalized in order to change their hip prosthesis at the hospital "la Croix-Rousse" in Lyon.
  Patients have to complete before the surgery a survey on occupational and environmental exposures to mineral dust.
  The prosthesis removed is composed by metal/polyethylene. It's a double mobility.
  The aim is to define the types of particles that cause the most tissue inflammation
  Groups: hip prosthesis metal/polyethylene in double mobility
Procedure: hip prosthesis removed ceramic/ polyethylene, simple mobility — Patients are hospitalized in order to change for their hip prosthesis at the hospital "la Croix-Rousse" in Lyon.
  Patients have to complete before the surgery a survey on occupational and environmental exposures to mineral dust.
  The prosthesis removed is composed by ceramic/polyethylene. It's a simple mobility.
  The aim is to define the types of particles that cause the most tissue inflammation
  Groups: hip prosthesis ceramic/polyethylene in simple mobility
Procedure: hip prosthesis removed ceramic/ polyethylene, double mobility — Patients are hospitalized in order to change their hip prosthesis at the hospital "la Croix-Rousse" in Lyon.
  Patients have to complete before the surgery a survey on occupational and environmental exposures to mineral dust.
  The prosthesis removed is composed by ceramic/polyethylene. It's a double mobility.
  The aim is to define the types of particles that cause the most tissue inflammation.
  Groups: hip prosthesis ceramic/polyethylene in double mobility
Procedure: Primary implanted hip prosthesis — Patients are hospitalized in order to have a first hip prosthesis at the hospital "la Croix-Rousse" in Lyon.
  Patients have to complete before the surgery a survey on occupational and environmental exposures to mineral dust.
  The patients will be received a first prosthesis.
  Groups: Primary implanted hip prosthesis
Procedure: hip prosthesis removed metal/metal — Patients are hospitalized in order to change their hip prosthesis at the hospital "la Croix-Rousse" in Lyon.
  Patients have to complete before the surgery a survey on occupational and environmental exposures to mineral dust.
  The prosthesis removed is composed by metal/metal. The aim is to define the types of particles that cause the most tissue inflammation
  Groups: metal / metal prosthesis removed
Procedure: hip prosthesis removed ceramic/ceramic — Patients are hospitalized in order to change their hip prosthesis at the hospital "la Croix-Rousse" in Lyon.
  Patients have to complete before the surgery a survey on occupational and environmental exposures to mineral dust.
  The prosthesis removed is composed by ceramic/ceramic. The aim is to define the types of particles that cause the most tissue inflammation
  Groups: ceramic / ceramic prosthesis removed

SUMMARY:
Hip arthroplasty is a treatment widely used in most inflammatory, traumatic and degenerative conditions of this joint. The longevity of implants may be disappointing in some cases, despite the promising results obtained during in vitro simulations. Early loco-regional or systemic dissemination, known since the 1990s, of wear particles from these prosthesis may reduce their life span.

The analysis of the particles in the synovial fluid and in the articular tissues by electron microscopy after digestion or directly by optical microscopy, will improve the knowledge on the mechanisms of wear.

This category 3 study is based on the case-control model and will be conducted in a national reference center (hospital la Croix-Rousse- Lyon). It will include a population of adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient,
* Patient including French,
* Patient witness: to be hospitalized in the orthopedic department of the Croix-Rousse hospital for a first hip prosthesis
* Patient test: to be hospitalized in the orthopedic department of the Croix-Rousse hospital for the removal of a hip prosthesis

Exclusion Criteria:

* Patient protected by law (guardianship, curatorship, safeguard of justice).
* Pregnant or lactating woman
* Patient with suspicion of infection on prosthesis
* Patient opposing his participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be having a surgery for the resumption of a hip prosthesis or for a first implantation
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-08-11 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
types of particles that cause the most tissue inflammation | day of surgery
  Types of wear particles most found in patients whose tissues are classified as inflammatory. The particles can be classified by size, shape, material and type of original prosthesis.

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Batailler, Dr, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Hôpital Edouard Herriot, Lyon
  - Hôpital de la Croix Rousse, Lyon